CLINICAL TRIAL: NCT03631771
Title: A Multicenter, Prospective Study to Evaluate the Risk of Hypothyroidism in Pediatric Patients Administered Intravascular Iohexol, Iodixanol, Iopromide, or Ioversol. THYROPED.
Brief Title: Pediatric Risk of Hypothyroidism With Iodinated Contrast Media
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: It was determined that a study is no longer required because the clinical question posed by the study has been answered through published literature
Sponsor: GE Healthcare (Industry)
Collaborators: Bayer (Industry); Guerbet/Liebel-Flarsheim (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GE-012-103/19476/OPY-44-002
Record Dates: First submitted 2018-08-13; First posted 2018-08-15 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Hypothyroidism
Keywords: Hypothyroidism; Child; Iodine; Iodinated contrast medium (ICM); Thyroid function test (TFT); Iodixanol; Iohexol; Iopromide; Ioversol
MeSH Terms: conditions — Hypothyroidism | interventions — Iohexol; iodixanol; iopromide; ioversol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Iodixanol, iohexol, iopromide, or ioversol (Experimental): Investigational medicinal product administered intravascularly per usual clinical practice at each participating institution. Doses will be per usual practice. The dose of ICM, timing of ICM administration in relation to the diagnostic procedure, rate of ICM administration, and route of ICM administration will be determined by the physician performing the enhanced radiologic procedure per medical need and local clinical practice.
  Interventions: Drug: Iohexol; Drug: Iodixanol; Drug: Iopromide; Drug: Ioversol

INTERVENTIONS:
Drug: Iohexol — Iohexol administered intravascularly
  Other Names: Omnipaque™
Drug: Iodixanol — Iodixanol administered intravascularly
  Other Names: Visipaque™
Drug: Iopromide — Iopromide administered intravascularly
  Other Names: Ultravist®
Drug: Ioversol — Ioversol administered intravascularly
  Other Names: Optiray®

SUMMARY:
This is a Phase 4 multicenter prospective study to estimate the proportion of patients aged birth to 3 years who develop hypothyroidism within 6 months after receiving intravascular iohexol (Omnipaque™), iodixanol (Visipaque™), iopromide (Ultravist®), or ioversol (Optiray®) as the iodinated contrast medium (ICM) for clinical evaluation during an ICM-enhanced diagnostic imaging procedure.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged birth to 3 years who, as part of the standard of care in the clinical practice of medicine, are referred to and will undergo a radiographic diagnostic imaging procedure that uses intravascularly administered iohexol (Omnipaque™), iodixanol (Visipaque™), iopromide (Ultravist®), or ioversol (Optiray®) as the ICM for contrast enhancement.
* Written informed consent has been given for the patient by one or more parents or other legally acceptable representatives, as required by local regulations and laws.
* When applicable (neonates), the patient's biological mother consents to providing information about her medical history and medication usage.
* The patient has normal pre-procedure (screening) serum TFTs (TSH, TT4, FT4, TT3), TSI, and urine (UI/UCr).
* The patient's pre-procedure (screening) serum chemistry is either normal or not clinically significantly abnormal.
* The patient has normal pre-procedure (screening) eGFR for age by the revised Schwartz formula [Schwartz et al 2009].
* The patient's parent(s) or other legally acceptable representative(s) is/are able and willing to comply with the study schedule and procedures.

Exclusion Criteria:

* The planned radiographic procedure is part of a clinical research study rather than clinical practice.
* The patient has known or suspected thyroid disease, Down syndrome (trisomy 21), or Type 1 diabetes.
* The patient currently receives thyroid hormone replacement therapy, or such therapy is planned or being considered.
* The patient has been exposed to thyroid protection for imaging procedures, within the last 6 months or such procedure is planned or being considered.
* The patient currently receives one or more anti-thyroid medications, or such therapy is planned or being considered.
* The patient has known or suspected past or present exposure to thyroid suppressants, including but not limited to drugs (e.g., amiodarone), inorganic iodide (potassium iodide, sodium iodide, etc.), perchlorate, thiocyanate, nitrate, lithium, and topical iodine disinfectant (e.g., povidone-iodine).
* The patient has undergone (or is expected to undergo during the study) radiation treatments to the head or neck.
* There is a high likelihood that the patient will undergo surgery or more than one ICM-enhanced procedure in the following 10 weeks.
* The patient has a history of hypersensitivity to ICM or any components, or a history of a severe cutaneous adverse reaction to ICM.

Max Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2022-03 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects who develop hypothyroidism post-ICM. | 6 months

SECONDARY OUTCOMES:
Proportion of subjects with changes from baseline in thyroid function tests that exceed the available literature-reported reference change values for these parameters (ca. >60% for TSH and >30% for thyroxine [T4]; [Chaler et al 2012]) | 6 months
Proportion of subjects with abnormal thyroid function tests at each time point. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul F. Sherwin, MD, PhD, Study Director — GE Healthcare; Zuzana Jirakova Trnkova, MD, PhD, Study Director — Bayer; Philippe Bourrinet, PharmD, Study Director — Guerbet